CLINICAL TRIAL: NCT00631618
Title: A Phase II Trial of Sutent in Metastatic Melanoma Patients With KIT Aberrations.
Brief Title: Clinical Trial of Sutent to Treat Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Pfizer (Industry); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, David Minor, MD, Medical Doctor, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA6181DN
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sunitinib

ARMS (1):
- Suntinib (Experimental): Suntinib
  Interventions: Drug: Sutent (sunitinib)

INTERVENTIONS:
Drug: Sutent (sunitinib) — The initial dose will be 50mg daily taken for 4 consecutive weeks followed by 2-weeks off to comprise a complete cycle of 6 weeks.
  Other Names: sunitinib malate

SUMMARY:
The purpose of this study is to investigate whether an investigational drug called sunitinib malate is safe and effective in treating metastatic melanoma in patients with KIT mutations.

KIT is a gene that "codes for" (contains the genetic code that the body uses to make) a protein on the surface of cells in your body that is important in cell growth and cell division. The KIT protein seems to play a role in abnormal cell growth seen in acute leukemia, germ cell tumors, gastrointestinal stromal tumors (GIST), and certain melanomas. Melanomas that arise on acral skin (palms, soles, nail beds), mucosal membranes, and chronically sun damaged skin have recently been found to frequently contain mutations or increased copy numbers of the KIT gene. Your tumor tissue has previously been tested and has been found to contain abnormalities in the KIT gene.

Sunitinib malate is drug that has been shown to inhibit the activity of the KIT protein. The FDA approved sunitinib in 2006 for patients with GIST. It has been shown that sunitinib malate works in these patients because of its activity against the KIT protein. The FDA also approved Sunitinib malate in 2006 for the treatment of metastatic kidney cancer, where its effectiveness is probably due to its ability to block a different set of proteins.

Sunitinib malate has not been approved by the FDA for the treatment of metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced stage III or IV melanoma with primary origin in mucosal, acral-lentiginous, or chronic sun-damaged skin. Advanced disease is defined as locally recurrent disease or metastatic disease not amenable to surgical therapy. Patients may enter tumor-testing phase even if they do not have recurrent disease.
* Aberration of the KIT gene or KIT receptor on in-vitro testing of their tumor tissue.
* Evidence of measurable disease by RECIST criteria [Appendix 2]. Bone lesions, ascites, peritoneal carcinomatosis or miliary lesions, pleural or pericardial effusions, lymphangitis of the skin or lung, cystic lesions, or irradiated lesions are not considered measurable.
* Resolution of all acute toxic effects of prior chemotherapy, immunotherapy, radiotherapy or surgical procedures to NCI CTCAE Version 3.0 grade ≤1.
* Adequate organ function
* ECOG performance status 0 or 1.

Exclusion Criteria:

* Major surgery or radiation therapy within 2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* NCI CTCAE Version 3.0 grade 3 hemorrhage within 4 weeks of starting the study treatment.
* Diagnosis of any second malignancy within the last 2 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, localized prostate cancer, or in situ cervical cancer.
* Active brain metastases, spinal cord compression, or evidence of symptomatic brain or leptomeningeal carcinomatosis on screening CT or MRI scan. Patients who have had central nervous system metastases treated by surgery or radiation therapy and with those CNS metastases considered in control will be eligible, provided measurable disease outside the CNS is present.
* Any of the following within the 2 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade > 2.
* Prolonged QTc interval on baseline EKG (>450 msec for males or >470 msec for females)
* Uncontrolled hypertension (> 160/100 mm hg despite optimal medical therapy).
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g., QOL, are allowed.
* Ongoing treatment with therapeutic doses of warfarin (low dose warfarin up to 2 mg po daily for thromboprophylaxis is allowed).
* Pregnant or breastfeeding.
* Life expectancy less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Determine the objective response rate of metastatic melanoma patients with KIT aberrations to therapy with sunitinib. | 5 years

SECONDARY OUTCOMES:
Study the safety and toxicity of sunitinib when given to metastatic melanoma patients with KIT aberrations. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David R Minor, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

REFERENCES:
- [Result] Minor DR, Kashani-Sabet M, Garrido M, O'Day SJ, Hamid O, Bastian BC. Sunitinib therapy for melanoma patients with KIT mutations. Clin Cancer Res. 2012 Mar 1;18(5):1457-63. doi: 10.1158/1078-0432.CCR-11-1987. Epub 2012 Jan 18. PMID 22261812